CLINICAL TRIAL: NCT00399932
Title: Non-invasive Evaluation of Hepatic Fibrosis in Patients With the Metabolic Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Prof Y Horsmans, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Other Study IDs: ELASTO1
Record Dates: First submitted 2006-11-14; First posted 2006-11-15 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Metabolic Syndrome
Keywords: metabolic syndrome; insulin resistance; NASH; hepatic fibrosis; Fibroscan; elastography by MRI
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — liver biopsy serum
Oversight: Data Monitoring Committee: No

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is now recognised as the hepatic complication of the metabolic syndrome of insulin resistance. In some patients, the disease can progress into steatohepatitis (NASH) which associates fatty liver, hepatocellular damage, chronic inflammation and variable and progressive fibrosis. The latter can evolve into cirrhosis and end-stage liver disease.

Thus the presence of fibrosis sign the severity of the disease, and therefore its accurate detection is crucial for the identification of patients in need of treatment and appropriate follow-up.

To date, histological examination of a biopsy of the liver is the gold standard in the diagnosis of fibrosis. the procedure is however associated with significant complication in 0.01 to 0.1% of cases and with sampling errors because it analyses only a minimal portion fo the liver.

The aim of the study is to evaluate, in a population of patients with the metabolic syndrome, whether non-invasive tests may identify those with hepatic fibrosis.

At inclusion, serum tests, fibroscan (elastography of the liver by ultra-sounds) and elastography by MRI will be performed. Those tests will be repeated within 2 months.

A liver biopsy will be performed if 2 out of the 3 (serum test, fibroscan or elastography) tests are suggestive of hepatic fibrosis.

This study will allow to determine

* whether hepatic fibrosis may be detected by non-invasive means in patients with NAFLD/NASH.
* whether there is a correlation between non-invase tests and liver biopsy for assessment of fibrosis and it severity
* whether the presence of fatty liver interfere with the results of the fibroscan and the elastography.
* whether there are metabolic factors associated with an increased risk of fibrosis in this population.

ELIGIBILITY:
Inclusion Criteria:

* metabolic syndrome with 3 out of 5 criteria (ATP III definition)

Exclusion Criteria:

* alcohol intake > 20g/day (women), > 30g/day (men)
* chronic liver disease of other cause: viral hepatitis (HBV, HCV), Wilson's disease, haemochromatosis, alpha1 anti-trypsin deficiency, drug-induced, ...
* decompensated cirrhosis (Child-Pugh 3)
* body weight > 120 Kg

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with type 2 diabetes
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2006-03; Primary Completion 2009-05 (Actual); Study Completion 2010-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yves J Horsmans, M.D.,PhD, Study Director — StLuc university hospital, Université catholique de Louvain (UCL), Brussels, Belgium
Locations (1):
- StLuc University Hospital, Brussels, Belgium